CLINICAL TRIAL: NCT02566733
Title: Performance of the Minto Model in Effect Site Mode for Target Controlled Infusion of Remifentanil During Cardiopulmonary Bypass
Brief Title: Minto Model in Effect Site Mode for Target-Controlled Infusion of Remifentanil During Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Remifentanil_CPB
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Anesthetics, Intravenous; Pharmacology; Anesthetics; Cardiopulmonary Bypass
Keywords: remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remiva (Experimental): This experimental group will use a generic drug of remifentanil, Remiva™ from Hana Pharmaceutical company.
  Interventions: Drug: Remiva
- Ultiva (Active Comparator): This arm group will use a brand-named drug of remifentanil, Ultiva™ from GlaxoSmithKline company.
  Interventions: Drug: Ultiva

INTERVENTIONS:
Drug: Remiva — Target controlled infusion of remifentanil (generic drug, Remiva™)
  Other Names: generic drug of remifentanil, Remiva™
  Arms: Remiva
Drug: Ultiva — Target controlled infusion of remifentanil (brand-named drug, Ultiva™)
  Other Names: brand-named drug of remifentanil, Ultiva™
  Arms: Ultiva

SUMMARY:
Target controlled infusion with remifentanil is widely used during cardiac surgery, wich is performed using the Minto model. It was derived from patients undergoing general surgery. However, pharmacokinetics of remifentanil can be changed during cardiopulmonary bypass. The investigators tested whether Minto model for target controlled infusion produces constant plasma remifentanil concentration during the cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with the ASA class I~III undergoing elective cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* Patients not using target controlled infusion during the operation
* Patients with drug/substance abuse
* Patients using analgesics before this study starts
* Pregnant women
* Patients who rejected study participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Median prediction error | during CPB

SECONDARY OUTCOMES:
changes of measured total remifentanil concentration | 1 hour after anesthesia induction, 30/60/90 min after the beginning of cardiopulmonary bypass, 1 hour after the end of cardiopulmonary bypass
Median absolute prediction error | during CPB

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea